CLINICAL TRIAL: NCT03889769
Title: Evaluation of Accuracy of One-Step Nucleic Acid Amplification (OSNA) in Diagnosis of Lymph Node Metastases of Papillary Thyroid Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Fabio Medas, Research fellow, University of Cagliari
Other Study IDs: NP20164594
Record Dates: First submitted 2019-03-23; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Papillary Thyroid Cancer; Lymph Node Metastases
MeSH Terms: conditions — Thyroid Cancer, Papillary; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: OSNA test — Analysis of lymph node with OSNA

SUMMARY:
The incidence of node metastases in papillary thyroid carcinoma (PTC) is high, ranging from 20% to 90%. Prophylactic central lymph node compartment dissection (CLND), suggested from the latest guidelines for high-risk tumors, meets resistance due to the high incidence of postoperative complications. Recently, new molecular biologic techniques, such as One Step Nucleic Acid Amplification (OSNA), have spread widely, allowing to quickly isolate, amplify and quantify mRNA encoding for proteins selectively present in neoplastic cells, as Cytokeratine-19. The aim of this study is to evaluate the application of OSNA to intraoperative diagnosis of node metastases of PTC.

DETAILED DESCRIPTION:
Papillary thyroid carcinoma (PTC) is the most common malignant thyroid neoplasm; it originates from follicular cells of thyroid gland, and represents over 80% of thyroid tumors. The incidence of PTC has progressively been increasing in the last decades, doubling since the 1970s, due to the diffusion of screening ultrasound. Although PTCs are considered slow-growing tumors, the incidence of node metastases is high, ranging from 20% to 90%. The real impact of node metastases on prognosis is still a matter of debate: reports in literature demonstrate a reduction of disease-free survival but are divergent on overall survival. Diagnostic tools have poor accuracy for central lymph node compartment, which is the most frequent site of metastases.

The last guidelines suggest a prophylactic central lymph node compartment dissection (CLND) in patients with high-risk PTC; nevertheless, this indication meets resistance due to the higher incidence of postoperative complications, especially hypoparathyroidism and recurrent laryngeal nerve (RLN) palsy.

Recently, new molecular biologic techniques have spread widely, mainly in diagnosis of node metastases in breast carcinoma; these assays allow to quickly isolate, amplify and quantify mRNA encoding for proteins selectively present in neoplastic cells, as Cytokeratine-19 (CK-19). One Step Nucleic Acid Amplification (OSNA) is routinely used in diagnosis of node metastasis in sentinel lymph node (SNL) of patients affected from breast cancer. The aim of this study is to evaluate if application of OSNA to intraoperative diagnosis of node metastases of PTC is possible.

ELIGIBILITY:
Inclusion Criteria:

Preoperative diagnosis of thyroid carcinoma

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with preoperative cytological diagnosis of papillary thyroid carcinoma (Tir4-Tir5)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-12-20 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of OSNA | 1 day
  Measurement of OSNA accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Giorgio Calò, Principal Investigator — University of Cagliari
Locations (1):
- Policlinico di Monserrato, Monserrato, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: Undecided